CLINICAL TRIAL: NCT00661349
Title: Prospective, Open Label and Randomized Clinical Trial About Hepatic Security of Antiretroviral Treatment Based on Kaletra Versus Nevirapine in Co-infected HIV/HCV Patients
Brief Title: Trial About Hepatic Security of Antiretroviral Treatment Based on Kaletra Versus Nevirapine in Co-infected HIV/HCV Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It has been impossible to achieve the number of patients defined by protocol
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A10-174 (KANELA)
Record Dates: First submitted 2008-04-10; First posted 2008-04-18 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Kaletra; Nevirapina; HCV chronic infection; Fibroscan; hepatic fibrosis; treatment experienced
MeSH Terms: conditions — HIV Infections; Liver Cirrhosis | interventions — Lopinavir; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nevirapine
  Interventions: Drug: Nevirapine
- 2 (Experimental): Lopinavir/ritonavir
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir — 2 ITIAN (o 1 ITIAN+TDF)+ lopinavir/ritonavir, 2 tablet 200/50 mg to 12 hours
  Arms: 2
Drug: Nevirapine — 2 ITIAN (o 1 ITIAN+TDF)+ nevirapine, 2 tablet 200/50 mg to 12 hours
  Arms: 1

SUMMARY:
In retrospective studies, acceleration of hepatic fibrosis has been seen in Nevirapine (NVP) treatment when compared with Protease Inhibitors (PI) boosted with ritonavir treatment in patients with Human Immunodeficiency Virus (HIV) and Hepatitis C Virus (HCV) infection. The high incidence in our country of HIV-HCV co-infection, the availability of a new Kaletra (LPV/r) formulation (more convenient and better tolerated than soft capsules) as well as the possibility of analyzing hepatic fibrosis evolution in a fast and bloodless way, make attractive a study that, in a prospective way, could check the benefits of substituting NVP by LPV/r on hepatic fibrosis in this community.

DETAILED DESCRIPTION:
The prevalence of the HIV-HCV co-infection in Spain is one of the highest because both infections are strongly related to parenteral drugs use; so, from 61 to 69 % of HIV infected patients are also HCV infected.

Acute HCV infection is asymptomatic in 60 to 70% of cases, being the chronification the natural illness evolution. 20% of the patients will develop hepatic cirrhosis after 20 to 30 years of being infected by the HCV. In cirrhosis cases, the hepatocellular carcinoma appears in a rate of 2 to 4% per year, according to studies done with HCV mono-infected patients. Fibrosis progression depends basically on the duration of HCV infection and on the age of infection, but also on other factors, like gender (is faster in men), alcohol consumption (worst over 50 g per day) and HIV co-infection. Several epidemiologist studies have described the negative impact of HIV co-infection, accelerating the progression to cirrhosis and the hepatocarcinoma.

The Highly Active Antiretroviral Treatment (HAART) has a positive impact on survival on co-infected patients, although the three drug families used in HAART can cause hepatic toxicity in this group of patients. Hepatic toxicity appears in 5 to 20% of patients, being more serious and common, but not exclusive, in case of NVP treatment.

On their part, not all PI have the same hepatotoxic profile. An association between serious hepatotoxicity and ritonavir at full strength, indinavir and indinavir plus saquinavir boosted with ritonavir has been found.

As far as fibrosis is concerned, there are studies that show that in HIV/HCV co-infected patients PI-based regimens are associated with a lower progression to fibrosis, while the progression rate to cirrhosis is higher in NVP-based regimens, mainly in those patients with advanced hepatic fibrosis.

Hepatic biopsy is considered the reference test to assess hepatic fibrosis, nevertheless it is an invasive, painful and with a low but potentially serious risk for the patient's life. Moreover, the viability of a hepatic biopsy can be doubted due to sampling error or interobservation variability. For that reason, several biochemist tests have been developed to reflect the hepatic fibrosis extent or stage in a reliable way. Recently a hepatic rigidity measure through elastography has been presented as a non-invasive and very promising method to assess hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or elder.
2. HCV and HIV co-infected patients.
3. Patients with antiretroviral treatment based in NVP plus 2 NRTIs (or 1 NRTI and Tenofovir), with undetectable viral load (under 50 copies/mL) during at least the last 24 weeks.
4. If women and of childbearing age, negative pregnancy test. Furthermore, barrier contraceptive method must be undertaken during the study.
5. Date and signature of the informed consent.

Exclusion Criteria:

1. Concomitant treatment with drugs that can significantly interact with the study drugs.
2. Opportunistic infections in the last 6 months.
3. Patients who can be candidates for an HCV infection treatment in the next 3 years.
4. Patients in who efficacy of previous NRTIs can not be ensured. For example, patients with mono or dual therapy history or with previous blips in whom NRTI-related mutations were identified that could reduce the sensibility to the used backbone.
5. Active alcohol consumption (over 50 g per day) or other substance abuse.
6. Pregnant or breastfeeding women.
7. Patients with transaminase level over 5 times the Upper Limit of Normality (ULN) or Creatinin over 2 mg/dL or Total Bilirubin over 3 times the ULN.
8. Any formal contraindication for being treated with the study drugs.
9. Patients who, basing in their antiretroviral treatment history, could be considered as being infected with a virus that has no sensibility to LPV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The average of hepatic rigidity increase in each group. Hepatic rigidity will be measured in kilopascals through elastography (Fibroscan). Distribution of hepatic rigidity will be normalized by a logarithmic transformat | From Basal to 144 week (last visit) every 3 months

SECONDARY OUTCOMES:
Virological and immunologic efficacy will be assessed through the proportion of patients with virological failure during the follow-up and the CD4 lymphocytes count of both treatment regimens. | From Basal to 144 week (last visit) every 3 months
The effect of both treatments in lipidic and glucidic metabolism will be assessed through the following variables: Total Cholesterol, HDL and LDL Cholesterol, Triglycerides and Glucose. | From Basal to 144 week (last visit) every 3 months
Higher than log 7.2 Kpa in patients with non-significant basal fibrosis (less than log 7.2 Kpa) | From Basal to 144 week (last visit) every 3 months
The security of each regimen will be studied through the proportion of patients who give up treatment because of adverse events and hepatic-related adverse events presence. | From Basal to 144 week (last visit) every 3 months
Toxicity will be determined depending on: Clinical History and Physical Examination; Coagulation, hemogram and chemistry tests, which will include: transaminase levels, GGT, alkaline phosphatase, bilirrubin, albumin, urea and creatinin | From Basal to 144 week (last visit) every 3 months
Mortality rate during the study will be evaluated. | From Basal to 144 week (last visit) every 3 months

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - H.U. Germans Trias i Pujol - Unitat VIH, Fundació Lluita contra la Sida, Badalona, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario de Valme, Seville